CLINICAL TRIAL: NCT06187324
Title: Accuracy of Host-derived Biomarkers in Diagnosing Symptomatic and Asymptomatic Apical Periodontitis and Predicting the Outcome of Endodontic Treatment: Controlled Clinical Trial
Brief Title: Accuracy of Host-derived Biomarkers in Diagnosing Symptomatic and Asymptomatic Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Zeena Tariq Abdulhadi, assistant professor, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: biomarkers in GCF
Record Dates: First submitted 2023-11-21; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Biomarkers
MeSH Terms: interventions — Environmental Biomarkers

STUDY DESIGN:
Intervention Model Description: two groups comparison,symptomatic and asymptomatic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- periopaper (Experimental): periopaper used to collect GCF
  Interventions: Diagnostic Test: biomarkers

INTERVENTIONS:
Diagnostic Test: biomarkers — by th use of perio paper GCF was collected and Biomarkers level was estimated

SUMMARY:
Apical lesions usually present clinically as a chronic infection, remaining as asymptomatic apical periodontitis(AAP). Because the balance among inflammation and bacteria is a dynamic process, AAP may undergo an acute exacerbation and become symptomatic, presenting as symptomatic apical periodontitis or acute abscess, or it may evolve from the acute to the chronic stage. Identification of specific biomarker could help in establishing more accurate diagnosis. Biological marker serves as a parameter that is indicative of underlying physiology and health of the tissue. It is measurable as well as quantifiable. The aim of this study: To assess the level of potential biomarkers in asymptomatic and symptomatic apical Periodontitis, and to determine the prediction potential of the same biomarkers for the outcome of endodontic treatment after 1year recall…

DETAILED DESCRIPTION:
Participants will be selected from patients attending the Restorative and Aesthetic Department in the College of Dentistry University of Baghdad. Consent form will be assigned with all participants prior to the study to take their agreement for participation. Also case sheet including all diagnostic procedures will be prepared and used with all cases. The involved tooth should not have more than 3 surfaces affected with caries including mesioocclusal(M0), distoocclusal(DO) or mesio occlusodistal( MOD). Cone beam computed tomography (CBCT) will be taken for the accused teeth. Gingival crevicular fluid(GCF) samples will be collected from the gingival sulcus of the test and healthy teeth within the same participant. The GCF samples will be centrifuged at 400-500 g for 4-5 min and Concentrations of Matrix metaloproteinases(MMP8), Tissue inhibitor(TIMP1),receptor activator of nuclear factor kappa-B(RANK), RANK ligand(RANKL) andosteoprotegerin( OPG) will be determined using ELISA test.

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy individuals with healthy periodontal status which can be detected by periodontal probing depth (PPD) and bleeding on probing (BOP).
* Both sexes and ages between 25-45 years old will be targeted.
* Patients with one or more SAP or AAP teeth will be included within this study.
* The involved tooth or teeth have to be one or both of the maxillary premolars either In one or both sides.
* Selected SAP and AAP has to be without periodontal diseases.

Exclusion Criteria:

Systematically unhealthy individuals or those who consumed any treatment that may affect periodontal condition.

* Consumption of antibiotics within 3-months prior to the study first examination.
* Periodontitis.
* Smoker.
* Pregnancy and lactation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Assessment the level of host-derived biomarkers (RANK,RANKL,OPG,MMP8,TIMP1)in asymptomatic and symptomatic apical periodontitis and their ability to predict the outcome of endodontic treatment: controlled clinical trial | 1 year
  mesearing level of biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sarhang Hama, PHD, Study Director — University of Sulaymania
Locations (1):
- Zeena, Baghdad, Iraq